CLINICAL TRIAL: NCT06342843
Title: Direct Superior Approach Versus PosteroLateral Approach in Total Hip Arthroplasty: a Multicenter Double Blinded Randomized Controlled Trial
Brief Title: Direct Superior Approach Versus PosteroLateral Approach in Total Hip Arthroplasty (SPLAsH)
Acronym: SPLAsH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Roelina Munnik, PhD, Researcher, Isala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPLAsH; NL81395.075.22 (Other: CCMO)
Record Dates: First submitted 2024-02-28; First posted 2024-04-02 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Intervention Model Description: multicenter, prospective, double blinded, randomized controlled intervention study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Posterolateral approach (PLA) (Active Comparator): THA by using the posterolateral approach
  Interventions: Procedure: Total Hip Arthroplasty
- Direct superior approach (DSA) (Active Comparator): THA using the direct superior approach
  Interventions: Procedure: Total Hip Arthroplasty

INTERVENTIONS:
Procedure: Total Hip Arthroplasty — a surgical procedure in which an orthopaedic surgeon removes the damaged bone and cartilage and replaces this with prosthetic components.

SUMMARY:
This study will compare postoperative pain, health related quality of life (HRQoL), function, rehabilitation, urinary incontinence, muscle atrophy and component positioning in total hip arthroplasty (THA) using the posterolateral approach (PLA) or the direct superior approach (DSA). In addition, the CT images will be used to validate a new metal artefact reduction technique.

DETAILED DESCRIPTION:
Objective: The primary objective is to evaluate health related quality of life (HRQoL) after THA using the DSA compared to the golden standard PLA in patients with incapacitating hip osteoarthritis after two weeks. The secondary objectives are divided into 1) long-term HRQoL evaluation, 2) physical performance, 3) radiologic muscle atrophy and component placement of the THA, 4) validation of a new metal artifact reduction technique for CT, and 5) relationship urinary incontinence and muscle atrophy.

Study design: Multicenter, prospective, double blinded, randomized controlled intervention study in which the used operation method is not shared with the patient until one year after surgery and in which the study researcher is also blinded.

Study population: A total of 211 men and women, age ≥ 18 years, with symptomatic hip osteoarthritis in whom THA is indicated.

Intervention (if applicable): For this randomized controlled trial (RCT), patients will be randomly allocated in one of two groups: one group receives THA by using PLA, the other group receives THA by using DSA.

Main study parameters/endpoints: As primary outcome specifically the Hip Disability and Osteoarthritis Outcome Score- Physical Function Short Form (HOOS-PS) is used for the short-term HRQoL.

Secondary parameters/endpoints are split up into different categories. 1) HRQoL evaluation on the long term using patient reported outcome measures (PROMs) (NRS score, Short form-12 (SF-12), HOOS subscales, Global rating of change, and Euro Quality of Life questionnaire). 2) Physical function using physical functioning test (Timed Up and Go test, 40-meter self-paced walk test for hip osteoarthritis and Stair Climb Test). 3) Muscle atrophy measurements using CT scans. Muscle atrophy is expressed in both quantity of muscle volume loss and extend of fatty infiltration using the Goutallier scale. Component placement is measured in different angles. 4) Evaluation of a new metal artifact reduction technique for CT images. 5) Relationship between muscle atrophy and urinary incontinence after total hip replacement.

Other study parameters include preoperative demographics such as age and gender, perioperative data such as blood loss, use of analgetics, operation time and postoperative complications such as infection, aseptic loosening and dislocation.

ELIGIBILITY:
Inclusion Criteria:

Subject

* Has symptomatic incapacitating coxarthrosis in whom total hip arthroplasty (THA) is indicated, diagnosed by both physical examination and pelvic/hip X-ray
* Has signed informed consent
* Is ageing 18 years or older at time of study entry
* Is competent and able to participate in follow-up

Exclusion Criteria:

* Previous ipsilateral hip surgery
* BMI >35 kg/m2
* Contralateral incapacitating coxarthrosis, diagnosed by both physical examination and pelvic/hip X-ray
* Neurological conditions influencing walking pattern
* Inability to walk without walking aid preoperatively
* Rheumatoid arthritis (RA)
* Severe hip dysplasia
* Cognitive impairment
* Malignancies or metastases involving the hip joint or the nearby soft tissues
* Inability to speak and write Dutch language

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Hip disability and Osteoarthritis Outcome Score - Physical Function Short Form | pre-operatively and 2 weeks, 6 weeks, 3months and 12 months postoperatively
  Evaluation symptoms and shortcomings in patients with hip complaints, 0-100 points, in which a higher score indicates less complaints

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) | pre-operatively and 2 weeks, 6 weeks, 3 months and 12 months postoperatively
  Pain scoring on a 10-point Likert scale: 0 no pain to 10 worst thinkable pain
Short Form-12 (SF-12) | pre-operatively and 2 weeks, 6 weeks and 12 months postoperatively
  general health status, scored on 101-point Likert scale, 0 being worst health to 100 being ideal health
Hip disability and Osteoarthritis Outcome Score (HOOS) | pre-operatively and 2 weeks, 6 weeks and 12 months postoperatively
  evaluates symptoms and shortcomings in patients with hip complaints 5-point Likert scale, in which a higher score means less symptoms
Euro Quality of Life (EQ-5D) | pre-operatively and 2 weeks, 6 weeks, 3 months and 12 months postoperatively
  measures health-related quality of life using 5 domains, questions scored on a 0-100 scale, the higher the score the better the quality of life
Global Rating of Change scale | pre-operatively and 2 weeks, 6 weeks, 3 months and 12 months postoperatively
  measures whether patient has improved or deteriorated over time to determine an effect of an intervention. It asks patients to assess their current health status compared to a previous time-point. 7 numerical values ranging from 7 (very much better) to 1 (very much worse)
Timed Up and Go test (TUG test) | pre-operatively and 2 weeks, 6 weeks and 12 months postoperatively
  measures time it takes for an individual to stand up from an armchair, walk a distance of 3 meters, turn around, walk back and sit down. the quicker the better.
40 meter self-paced walk test for hip osteoarthritis | pre-operatively and 2 weeks, 6 weeks and 12 months postoperatively
  assesses the time it takes to walk 40 meters in patients with hip or knee osteoarthritis
Stair climb test | pre-operatively and 2 weeks, 6 weeks and 12 months postoperatively
  measures the time an individual needs to ascend and descent a stair with 10 steps
Muscle atrophy by using Computer Tomography (CT) scanner | pre-operatively and 12 months postoperatively
  Muscular atrophy of the short external rotator muscles will be measured absolutely in cm^3 using the Tumor Tracking Tool of Philip IntelliSpace Portal, version 9.0.
Computer Tomography (CT) image with orthopedic metal artefact reduction (O-MAR) | pre-operatively and 12 months postoperatively
  Computer Tomography (CT) image of the pelvis and some slices at the height of the knee condyles. The scans will be reconstructed with a slice thickness of 0.9 of 1 mm and with an additional soft tissue filter. The pre-operative CT scans will be performed with a kilovoltage peak (kVp) of 120. The post-operative scans will be performed at 140 kVp, which helps to mitigate metal artifacts. In addition, the post-operative CT scans will be edited with metal artefact reduction for orthopedic implants (O-MAR; Philips Healthcare). All CT scans will be analyzed on a 23.8-inch Liquid-crystal display (LCD) monitor with a resolution of 1920x1080 pixels.
Postoperative cup position on Computer Tomography (CT) image | 12 months postoperatively
  The initial abduction/inclination of the cup, angle α, is measured on a coronal Computer Tomography (CT) image with respect to the ischial bone, which is used as internal reference. The anterior opening angle of the cup (angle β) is measured on the axial slice at the middle of the head of the prosthesis in which the posterior acetabulum is used as an internal reference. The angle of the neck of the prosthesis relative to the horizontal plane, angle a, is measured in the coronal slice containing the thickest diameter of the neck and is also measured with respect to the ischial bone. The anteversion angle of the neck around the vertical axis, angle b, is measured in the axial slice containing the greatest diameter of the neck with respect to the posterior acetabulum.
Comparing definite cup position with preoperative planned cup position | pre- operatively and 12 months postoperatively
  The initial abduction/inclination of the cup, angle α, is measured with respect to ischial bone, which is used as internal reference. The anterior opening angle of cup (angle β) is measured on axial slice at the middle of the head of the prosthesis in which the posterior acetabulum is used as internal reference. The angle of the neck of the prosthesis relative to the horizontal plane, angle a, is measured in coronal slice containing the thickest diameter of the neck and is measured with respect to ischial bone. The anteversion angle of the neck around the vertical axis, angle b, is measured in the axial slice Pre-operative hip component planning will be conducted using X-ray and CT images. Regarding component planning, the use of X-ray is sufficient. 3D planning using CT images will be performed retrospectively. Cup position will be compared between the 2D and 3D planning and with the definite positions
Comparing definite component position with surgeon's perioperative estimation of component position | direct postoperative and 12 months postoperatively
  The surgeon writes a report of the performed procedure in which the estimated and targeted degrees inclination of the cup and degrees anteversion of the cup and stem are noted. Results will be compared to the component positions as measured on the postoperative CT scan.
  The initial abduction/inclination of the cup, angle α, is measured with respect to ischial bone, which is used as internal reference. The anterior opening angle of the cup (angle β) is measured on the axial slice at the middle of the head of the prosthesis in which posterior acetabulum is used as an internal reference. The angle of the neck of the prosthesis relative to the horizontal plane, angle a, is measured in the coronal slice containing the thickest diameter of the neck and is also measured with respect to the ischial bone. The anteversion angle of the neck around the vertical axis, angle b, is measured in the axial slice containing the greatest diameter of the neck with respect to the posterior acetabulum.
overall image quality | pre- operatively and 12 months postoperatively
  Images will be edited by deep-learning metal artifact reduction technique (DL-MAR) and by O-MAR. The post-surgery images with and without O-MAR and the images with DL-MAR will be scored by four radiologists. During this assessment, the radiologist will also have access to the pre-surgery Computer Tomography (CT) scans. The images with and without O-MAR and with DL-MAR will be scored by the radiologists using a five-point scale. The images will be scored on: overall image quality. A five point scale with score 1-5 will be used, including very poor (1), poor (2), fair (3), good (4) and excellent (5).
image diagnostic confidence | pre- operatively and 12 months postoperatively
  Images will be edited by deep-learning metal artifact reduction technique (DL-MAR) and by O-MAR. The post-surgery images with and without O-MAR and the images with DL-MAR will be scored by four radiologists. During this assessment, the radiologist will also have access to the pre-surgery Computer Tomography (CT) scans. The images with and without O-MAR and with DL-MAR will be scored by the radiologists using a five-point scale. The images will be scored on: 1) diagnostic confidence for bone, 2) diagnostic confidence for muscle, 3) diagnostic confidence for pelvic organs. a five point scale with score 1-5 will be used, including very poor (1), poor (2), fair (3), good (4) and excellent (5).
metal artifacts on images | pre- operatively and 12 months postoperatively
  Images will be edited by deep-learning metal artifact reduction technique (DL-MAR) and by O-MAR. The post-surgery images with and without O-MAR and the images with DL-MAR will be scored by four radiologists. During this assessment, the radiologist will also have access to the pre-surgery Computer Tomography (CT) scans. The images with and without O-MAR and with DL-MAR will be scored by the radiologists using a five-point scale. The images will be scored on: severity of metal artifacts. a five-point scale including severe (1), pronounced (2), moderate (3), mild (4) and none (5) will be used.
Incontinence Severity Index (ISI) | pre-operatively and 6 weeks and 12 months postoperatively
  this index consists of two questions about the frequency and the quantity of urinary incontinence (92). The value of each question will be multiplied. A higher score means more severe urinary incontinence.
Urinary Distress Inventory, Short Form (UDI-6) | pre-operatively and 6 weeks and 12 months postoperatively
  the UDI-6 consists of six items about the experiences with several symptoms and to what degree the patients bothers (93). A four-point Likert scale is used in the degree part (1 = not at all - 4 = greatly.). Total score is used as outcome. A higher total score means a higher disability.
Patient Global Impression of Severity (PGIS) | pre-operatively and 6 weeks and 12 months postoperatively
  one question about the severity of the urinary incontinence (94). A four-point Likert scale is used (1 = none - 4 = severe).
Incontinence Impact Questionnaire Short Form (IIQ-7) | pre-operatively and 6 weeks and 12 months postoperatively
  the IIQ-7 consists of seven items on the impact of urinary incontinence on activities, participation in daily life, social contacts and emotional status (93). A four-point Likert scale is used (1 = not at all - 4 = greatly.). A higher total score means a bigger impact.
Incontinence after Total Hip Arthroplasty | 6 weeks and 12 months postoperatively
  this customized question concerns the opinion of the subject if urinary incontinence is changed after the total hip arthroplasty. This question will only be administered at six weeks and one year postoperatively.participation in daily life, social contacts and emotional status (93). A four-point Likert scale is used (1 = not at all - 4 = greatly.). A higher total score means a bigger impact.

CONTACTS AND LOCATIONS:
Overall Officials: Harmen B. Ettema, MD/PhD, Principal Investigator — Isala
Locations (3):
- Netherlands (3):
  - Amphia, Breda, North Brabant
  - Isala, Zwolle, Overijssel
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland

IPD SHARING:
Plan to Share IPD: No